CLINICAL TRIAL: NCT04210908
Title: Ultrasound Imaging Biofeedback for Shortening the Second Stage of Labor: a Randomized Prospective Study
Brief Title: Biofeedback for Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Principal Investigator, Eran Brazilay, MD PhD, Head of the Obstetric and Gynecologic Ultrasound unit, Assuta Ashdod Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0064-19-AAA
Record Dates: First submitted 2019-12-15; First posted 2019-12-26 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Labor Long; Labour;Obstructed
Keywords: Biofeedback; Second stage of labor; Operative delivery; Transperineal ultrasound
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Intervention Model Description: Open label randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental): The patient will be instructed to bear down during 4 consecutive contractions while monitoring head descent using transperineal ultrasound. In the study group, patients will observe the descent of the head during contraction on the ultrasound display screen.
  Interventions: Other: Visual biofeedback
- Control (No Intervention): The patient will be instructed to bear down during 4 consecutive contractions while monitoring head descent using transperineal ultrasound. In the control group, patients will not observe the ultrasound display screen.

INTERVENTIONS:
Other: Visual biofeedback — Patient will observe the descent of the fetal head as they push during contractions
  Arms: Biofeedback

SUMMARY:
The purpose of this study is to examine whether transperineal ultrasound as visual biofeedback can be used during labor as an effective tool for shortening the second stage of labor and reducing the need for instrumental delivery, in a prospective randomized design.

DETAILED DESCRIPTION:
Biofeedback provides patients with better control of their body and their physiological reactions respective of the examined process, such as stress/anxiety, sports activity, labor, etc.

Women under epidural anesthesia, may frequently feel lack of control over the birthing process and difficulty in bearing down effectively, which is a very significant part of the second stage of labor.

Transperineal ultrasound during labor is a standard procedure in many medical centers in the world, mainly used to assist obstetricians in evaluating the progress of labor, fetal head position and assessing the chances of successful operative delivery. One of the most common tools used in transperineal ultrasound in measurement of the angle of progression, which has been suggested as a subjective method for assessing fetal station and for predicting successful vaginal delivery. A preliminary non-randomized study raised the possibility that the use of transperineal ultrasound during labor as a biofeedback tool may shorten the second stage of labor.

The purpose of this study is to examine whether this tool can be used during labor as an effective tool for shortening the second stage of labor and reducing the need for instrumental delivery, in a prospective randomized design.

ELIGIBILITY:
Inclusion Criteria:

1. First labor
2. Full dilation
3. Head position between SP-1 and SP+2.
4. Epidural anesthesia
5. No contraindication for vaginal delivery
6. Parturient informed consent

Exclusion Criteria:

1. Participation in parallel studies.
2. Category III fetal monitoring requiring immediate delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in delivery
Enrollment: 100 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Duration of the second stage of labor | Up to 6 hours
  Minutes from first documentation of full dilatation to delivery.

SECONDARY OUTCOMES:
Mode of delivery | Up to 6 hours
  Mode of delivery (categorical): spontaneous vaginal, operative vaginal or cesarean
Neonatal 1 minute Apgar score | Up to 6 hours
  Apgar score at 1 minute after delivery (scale of 0-10)
Neonatal 5 minute Apgar score | Up to 6 hours
  Apgar score at 5 minute after delivery (scale of 0-10)
Cord pH | Up to 6 hours
  Umbilical cord blood pH
Postpartum hemorrhage | Up to 24 hours
  Rate of early postpartum hemorrhage (during first 24 hours)
Maternal perineal tears | Up to 6 hours
  Maternal perineal tear grade (categorical): None and grades 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Eran Barzilay, MD PhD, Principal Investigator — Samson Assuta Ashdod University Hospital
Locations (1):
- Assuta Ashdod Hospital, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalache KD, Duckelmann AM, Michaelis SA, Lange J, Cichon G, Dudenhausen JW. Transperineal ultrasound imaging in prolonged second stage of labor with occipitoanterior presenting fetuses: how well does the 'angle of progression' predict the mode of delivery? Ultrasound Obstet Gynecol. 2009 Mar;33(3):326-30. doi: 10.1002/uog.6294. PMID 19224527
- [Background] Gilboa Y, Frenkel TI, Schlesinger Y, Rousseau S, Hamiel D, Achiron R, Perlman S. Visual biofeedback using transperineal ultrasound in second stage of labor. Ultrasound Obstet Gynecol. 2018 Jul;52(1):91-96. doi: 10.1002/uog.18962. Epub 2018 May 29. PMID 29155474
- [Background] Diegmann EK, Andrews CM, Niemczura CA. The length of the second stage of labor in uncomplicated, nulliparous African American and Puerto Rican women. J Midwifery Womens Health. 2000 Jan-Feb;45(1):67-71. doi: 10.1016/s1526-9523(99)00019-7. PMID 10772737
- [Background] Levy R, Zaks S, Ben-Arie A, Perlman S, Hagay Z, Vaisbuch E. Can angle of progression in pregnant women before onset of labor predict mode of delivery? Ultrasound Obstet Gynecol. 2012 Sep;40(3):332-7. doi: 10.1002/uog.11195. PMID 22605649